CLINICAL TRIAL: NCT03148613
Title: Carbon Monoxide Breath Sensor System (COBSS) Performance, Human Factors, and Usability Assessment in a Single Visit
Brief Title: Carbon Monoxide Breath Sensor System Performance, Human Factors, and Usability Assessment Conducted in a Single Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Utley, MD (Industry)
Collaborators: UserWise, LLC (Industry)
Responsible Party: Sponsor-Investigator, David Utley, MD, President and CEO, Pivot Health Technologies Inc.
Organization: Pivot Health Technologies Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CS-401
Record Dates: First submitted 2017-04-26; First posted 2017-05-11 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: All subjects experience device use compared to a control device (predicate).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 18-49 year old smokers using COBSS (Other): Younger smokers - Assessment of intended user performance in use scenarios, user documentation assessment, subjective feedback and rating scales.
  NOTE: 18-49 year Age Arm intended to evaluate human factors and usability of COBSS in younger smokers
  Interventions: Device: Carbon Monoxide Breath Sensor System (COBSS); Device: Bedfont - Micro+™ Smokerlyzer®
- ≥50 year old smokers using COBSS (Other): Older smokers- Assessment of intended user performance in use scenarios, user documentation assessment, subjective feedback and rating scales.
  NOTE:≥50 year Age Arm intended to evaluate human factors and usability of COBSS in younger smokers
  Interventions: Device: Carbon Monoxide Breath Sensor System (COBSS); Device: Bedfont - Micro+™ Smokerlyzer®

INTERVENTIONS:
Device: Carbon Monoxide Breath Sensor System (COBSS) — Carbon Monoxide Breath Sensor System (COBSS): Device to measure carbon monoxide levels in one's breath and inform the user.
Device: Bedfont - Micro+™ Smokerlyzer® — Bedfont - Micro+™ Smokerlyzer® : Predicate Device to measure carbon monoxide levels in one's breath.

SUMMARY:
Prospective, open label, single center clinical study enrolling 70 subjects to study Performance, Human Factors, and Usability for the Carbon Monoxide Breath Sensor System (COBBS)

DETAILED DESCRIPTION:
Performance:

* Non-invasively measure carbon monoxide (CO) levels in the exhaled breath of study subjects using two different types of measurement devices.
* Assess the correlation between the measured CO levels (in parts per million, or ppm) of the study CO breath sensor (Carrot Sense) and the predicate CO breath sensor (Bedfont).

Human Factors and Usability:

* Ensure that representative intended users are able to operate the COBSS independently.
* Validate appropriate mitigations of use related hazards identified in risk management documentation.
* Uncover previously unforeseen use errors.

NOTES:

* The study design allows for the assessment of a performance endpoint and human factors endpoint in a single study.
* Each participant will complete the study in a single visit which will include the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 90 minutes.

ELIGIBILITY:
Subject who self-report smoking 2 or more cigarettes each day

Inclusion Criteria:

* 18-80 years of age
* English speaking
* Owns and uses a smartphone
* Willing to sign the Informed Consent Form

Exclusion Criteria:

• Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Utley, MD, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Carrot Sense, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 18-49 Year Old Smokers Using COBSS: Younger smokers - Assessment of intended user performance in use scenarios, user documentation assessment, subjective feedback and rating scales.
  NOTE: 18-49 year Age Arm intended to evaluate human factors and usability of COBSS in younger smokers
  Carbon Monoxide Breath Sensor System (COBSS): Carbon Monoxide Breath Sensor System (COBSS): Device to measure carbon monoxide levels in one's breath and inform the user.
  Bedfont - Micro+™ Smokerlyzer®: Bedfont - Micro+™ Smokerlyzer® : Predicate Device to measure carbon monoxide levels in one's breath.
- ≥50 Year Old Smokers Using COBSS: Older smokers- Assessment of intended user performance in use scenarios, user documentation assessment, subjective feedback and rating scales.
  NOTE:≥50 year Age Arm intended to evaluate human factors and usability of COBSS in younger smokers
  Carbon Monoxide Breath Sensor System (COBSS): Carbon Monoxide Breath Sensor System (COBSS): Device to measure carbon monoxide levels in one's breath and inform the user.
  Bedfont - Micro+™ Smokerlyzer®: Bedfont - Micro+™ Smokerlyzer® : Predicate Device to measure carbon monoxide levels in one's breath.
Period: Overall Study
Arm/Group | 18-49 Year Old Smokers Using COBSS | ≥50 Year Old Smokers Using COBSS
Started | 39 | 31
Completed | 39 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18-49 Year Old Smokers Using COBSS | ≥50 Year Old Smokers Using COBSS | Total
Number analyzed (Participants) | 39 | 31 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 30 | 69
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 21 | 17 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 9 | 17
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 39 | 31 | 70
smoke frequency [Count of Participants; unit: Participants]
  1 per day | 2 | 0 | 2
  2 - 7 per day | 21 | 10 | 31
  8 or more per day | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Performance Variable - Correlation of Carbon Monoxide (CO) Measurements Between COBSS and Predicate Devices
Description: CO concentrations in parts per million (ppm) in exhaled breath from subjects at a single visit will be assessed and reported in order to compare the CO measurements from COBSS to a control (predicate) device. The correlation will be reported as an R value.
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 90 minutes.
  COBSS breath sample will take approximately 1 minute. Breath sample with the control device will take approximately 1 minute. The breath samples will be collected within 5-10 minutes of each other.
Time Frame: 1 minute
Population: The performance outcome was designed to evaluate all the participants together, thus the cohorts (arms/groups) were not evaluated separately for this outcome. The cohorts were used for the human factors and usability portion of the study, but are not applicable for this outcome.
  The R value reported is the correlation coefficient between 70 paired CO measurement values taken with the COBSS and predicate devices, by the 70 participants.
Measure: Number; unit: Correlation coefficient (R-value)
Groups:
- All Participants: Paired breath samples from each participant
  Carbon Monoxide Breath Sensor System (COBSS): Carbon Monoxide Breath Sensor System (COBSS): Device to measure carbon monoxide levels in one's breath and compared to predicate device
  Each participant measured carbon monoxide with both the COBSS and the predicate device. These CO measures were paired and used in a regression analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 70
Correlation coefficient (R-value) | 0.9878

2. Primary Outcome: Human Factors - User Performance in Use Scenarios Assessment With Observer Ratings
Description: User performance of participants in intended use scenarios will be assessed at a single visit. Participants will be observed if they can set up the device, use the device and interpret results. Observer ratings include 'Successful' and 'Unsuccessful'. Specific attention will be given to assess if any harms can occur from observed use errors. Outcome measure data table is tally of participants who were 'Successful' in each use scenario.
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 90 minutes.
  Observations are made throughout the study session. Assessments for individual tasks will take approximately 1 minute and assessments will be made over the study session which can last up to 90 minutes.
Time Frame: 1 minute for each question; up to 90 minutes for study session
Population: Outcome measure data table is tally of participants who were 'Successful' in each use scenario.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Carbon Monoxide Breath Sensor System (COBSS): Carbon Monoxide Breath Sensor System (COBSS): Device to measure carbon monoxide levels in one's breath and compared to predicate device
Arm/Group | 18-49 Year Old Smokers Using COBSS | ≥50 Year Old Smokers Using COBSS | All Participants
Number analyzed (Participants) | 39 | 31 | 70
Participants
  set up the device- Pair Breath Sensor | 34 | 25 | 59
  use the device - submit a breath sample | 37 | 29 | 66
  interpret results | 38 | 31 | 69

3. Secondary Outcome: User Documentation Assessment With Questionnaire With Observer Ratings
Description: Participant understanding of user documentation will be assessed at single visit. User documentation includes packaging information, quick start guide, reference card, and user manual. Observer ratings include 'Successful' and 'Unsuccessful'.
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 90 minutes.
  Observations are made throughout the study session. Assessments for individual tasks will take approximately 1 minute each. The User documentation assessment portion of the study session will last up to 30 minutes.
  The 5-Point Likert Scale for Clarity has the following answer options: 5 - Very Clear; 4 - Clear; 3 - Neither Clear nor Unclear; 2 - Unclear; and 1 - Very Unclear.
  Higher values of this scale represent a better outcome, which is greater clarity/understanding.
Time Frame: Up to 90 minutes
Population: How clear or unclear were the User Manual Reference Card, and Quick Start Guide?
Measure: Count of Participants; unit: Participants
Arm/Group | 18-49 Year Old Smokers Using COBSS | ≥50 Year Old Smokers Using COBSS | All Participants
Number analyzed (Participants) | 38 | 31 | 69
Participants
  5 - Very Clear | 23 | 17 | 40
  4 - Clear | 13 | 10 | 23
  3 - Neither Clear nor Unclear | 2 | 1 | 3
  2 - Unclear | 0 | 2 | 2
  1 - Very Unclear | 0 | 1 | 1

4. Secondary Outcome: Number of Participants Answering "No" for the Subjective Feedback With Questionnaire
Description: Subjective feedback focusing on any concerns (i.e. 'yes', 'no') on using device will be assessed at single visit.
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 90 minutes.
  *Row title truncated due to character limit. Actual question asked: Were there any points during this portion of the study that you experienced difficulty or had concerns about the product? Subjective feedback focusing on any concerns prior to the conclusion of the study session. Subjective feedback questions will take approximately 1-3 minutes each. The Subjective feedback portion of the study session will last up to 5 to 15 minutes.
Time Frame: Up to 90 minutes
Population: Outcome measure data table is tally of participants answering No.
Measure: Count of Participants; unit: Participants
Arm/Group | 18-49 Year Old Smokers Using COBSS | ≥50 Year Old Smokers Using COBSS | All Participants
Number analyzed (Participants) | 38 | 31 | 69
Participants
  Were there any points during ... that you experienced difficulty or had concerns about the product?* | 30 | 23 | 53
  Did you experience any moments of hesitation while using the product? | 33 | 27 | 60
  Did you have any safety concerns regarding the product or labeling? | 35 | 26 | 61

5. Secondary Outcome: Participant Assessment With Questionnaire Rating Scales
Description: Participant will be asked to provide ratings on the following:
  * How would you rate the ease or difficulty using the device and phone app? 5 - Very Clear; 4 - Clear; 3 - Neither Clear nor Unclear; 2 - Unclear; 1 - Very Unclear
  * How easy or difficult was it to understand and interpret the test results?
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 90 minutes.
  Participant will provide the ratings prior to the conclusion of the study session. Participant assessment with questionnaire rating scales will take approximately 1-2 minutes each. The Subjective feedback portion of the study session will last up to 5 minutes.
Time Frame: Up to 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 18-49 Year Old Smokers Using COBSS | ≥50 Year Old Smokers Using COBSS | All Participants
Number analyzed (Participants) | 38 | 31 | 69
Participants
  How would you rate the ease or difficulty using the device and phone app?: 5 - Very Easy | 26 | 8 | 34
  How would you rate the ease or difficulty using the device and phone app?: 4 - Easy | 9 | 18 | 27
  How would you rate the ease or difficulty using the device and phone app?: 3 - Neither easy nor difficult | 3 | 2 | 5
  How would you rate the ease or difficulty using the device and phone app?: 2 - Difficult | 0 | 2 | 2
  How would you rate the ease or difficulty using the device and phone app?: 1 - Very difficult | 0 | 1 | 1
  How easy or difficult was it to understand and interpret the test results?: 5 - Very Easy | 29 | 17 | 46
  How easy or difficult was it to understand and interpret the test results?: 4 - Easy | 8 | 10 | 18
  How easy or difficult was it to understand and interpret the test results?: 3 - Neither easy nor difficult | 1 | 2 | 3
  How easy or difficult was it to understand and interpret the test results?: 2 - Difficult | 0 | 2 | 2
  How easy or difficult was it to understand and interpret the test results?: 1 - Very difficult | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were observed for over the 90 minutes study session for each participant.
Arm/Group | 18-49 Year Old Smokers Using COBSS | ≥50 Year Old Smokers Using COBSS | All Participants
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/31 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/31 | 0/70
Other Adverse Events (participants affected / at risk) | 0/39 | 0/31 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT03148613/Prot_SAP_001.pdf